CLINICAL TRIAL: NCT00288795
Title: A Randomized Study of Polarity or Massage Therapy to Reduce Fatigue in Breast Cancer Patients During Radiation Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC U4104
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Fatigue
Keywords: Fatigue; Polarity; Massage
MeSH Terms: conditions — Fatigue | interventions — Massage

ARMS (3):
- 1 (No Intervention): Standard Care
- 2 (Other): Massage Treatment
  Interventions: Other: Massage Therapy
- 3 (Other): Polarity Treatment
  Interventions: Other: Polarity Therapy

INTERVENTIONS:
Other: Massage Therapy — Therapeutic Touch
  Arms: 2
Other: Polarity Therapy — Use of energy fields to alleviate distress and achieve balance in the body
  Arms: 3

SUMMARY:
This research study is being conducted to compare the effectiveness of two types of complimentary medicine treatments to see if they will reduce the fatigue experienced by breast cancer patients receiving radiation therapy. The treatments being studied are Polarity Therapy and Massage Therapy.

The primary study hypothesis is that Polarity Therapy will be efficacious in relieving fatigue in breast cancer patients receiving radiation treatments.

The secondary hypothesis is that Polarity Therapy will be efficacious in improving health-related quality of life in breast cancer patients receiving radiation treatments.

DETAILED DESCRIPTION:
This is a randomized three-arm clinical trial of an intervention examining the efficacy of Polarity Therapy for the relief of fatigue associated with radiation treatments in breast cancer patients. Patients who meets the eligibility criteria and who have signed the consent form will be randomized to one of three trial arms: 1) Polarity Treatment 2) Massage treatment 3) Standard Care. Three treatments will be administered in the 4th, 5th, and 6th calendar weeks of radiation treatment. There will be weekly blood draws to assess cytokine levels. In addition, 6 saliva samples will be gathered per day for 2 days during each of the 4 study weeks to assess cortisol levels. Saliva samples will be completed by the participant at home. An actigraph will be worn for the 28 day study period to assess activity and sleep. Patients randomized to the Standard Care Arm will receive a Polarity or Massage treatment gratis following the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Fatigue of 2 or greater on Symptom Inventory
* Received at least 8 radiation treatments
* Able to read English

Exclusion Criteria:

* Be receiving concurrent chemotherapy
* Have bone metastasizes
* Be taking methylphenidate, modafinil, sedatives, or anxiolytics
* Have a hemoglobin <11g/dL.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Fatigue: Brief Fatigue Inventory and the Multidimensional Fatigue Symptom Inventory; objectively via actigraphy; mood via the Fatigue/Inertia subscale of the Monopolar Profile of Mood States. | 4 wk

SECONDARY OUTCOMES:
Health -Related Quality of Life: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F). Quality of sleep assessed subjectively with Pittsburgh Sleep Quality Inventory and a Sleep Diary. | 4 wk

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mustian, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester James P. Wilmot Cancer Center, Rochester, New York, United States

REFERENCES:
- [Background] Mustian KM, Roscoe JA, Palesh OG, Sprod LK, Heckler CE, Peppone LJ, Usuki KY, Ling MN, Brasacchio RA, Morrow GR. Polarity Therapy for cancer-related fatigue in patients with breast cancer receiving radiation therapy: a randomized controlled pilot study. Integr Cancer Ther. 2011 Mar;10(1):27-37. doi: 10.1177/1534735410397044. Epub 2011 Mar 7. PMID 21382958